CLINICAL TRIAL: NCT01755169
Title: Ketamine in Chronic Kid's (KiCK) Pain
Acronym: KiCK Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to enroll sufficient patients
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Amy-Lee Bredlau, Director, Pediatric Brain Tumor Program, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KiCK Pain
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Child; Pediatric; Ketamine
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ketamine 0.25 mg/kg/dose (Experimental): A 5mL solution of 0.25 mg/kg/dose of ketamine will be given three times daily for 2 weeks.
  Interventions: Drug: Ketamine
- Ketamine 0.5 mg/kg/dose (Experimental): A 5mL solution of 0.5 mg/kg/dose of ketamine will be given three times daily for 2 weeks.
  Interventions: Drug: Ketamine
- Ketamine 1 mg/kg/dose (Experimental): A 5mL solution of 1 mg/kg/dose of ketamine will be given three times daily for 2 weeks.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Participants on active treatment are given ketamine orally for 2 weeks, at varying dosages (1 dosage per participant).
  Other Names: Ketalar
  Arms: Ketamine 0.25 mg/kg/dose; Ketamine 0.5 mg/kg/dose; Ketamine 1 mg/kg/dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to select the most tolerable dose of oral ketamine for children with chronic pain. Children will be given either placebo or one of three dosages of oral ketamine for 2 weeks. The dosage that is most tolerable will be selected for further study.

DETAILED DESCRIPTION:
Children with chronic pain are randomized to one of four arms (three study drug arms, one placebo arm) in a randomized, double-blinded fashion. Children are treated for 2 weeks and then monitored for an additional 12 weeks. Study participation is a total of 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject, parent, or guardian willing and able to give informed consent
* NRS for pain over the past 24 hours >4 at baseline
* Chronic pain, which has been present for >3 months, or persisting longer than is normal for the underlying diagnosis
* Chronic pain related to physiologic diagnoses including but not limited to: cancer, rheumatologic disease, sickle cell anemia, cystic fibrosis, pancreatitis, and neuromuscular disease (e.g. Duchenne muscular dystrophy)
* Able to tolerate and cooperate with neurocognitive assessment
* Age 8-20 years old

Exclusion Criteria:

* If they are known or suspected to have drug addiction
* Uncontrolled psychiatric disorder such as depression, schizophrenia, or bipolar disorder
* Uncontrolled hypertension
* Known liver disease or elevation of AST or ALT greater than 3 times the upper limit of normal.
* Previous intolerance or allergic reaction to ketamine
* Pregnancy
* Use of CYP3A4 inhibitors or inducers within the 2-week period prior the study drug administration or within 5 half-lives of the respective medication, whichever is longer, until study conclusion.
* Consumption of grapefruit or grapefruit products from at least 2 weeks prior to study drug administration until study conclusion.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy-Lee Bredlau, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 7 patients enrolled on the trial. However, 2 participants withdrew from the trial before they were randomized and 1 participant withdrew from the trial before being treated. Hence, the total number of patients for assessment is 4.
Groups:
- Placebo: Placebo
Period: Overall Study
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Placebo
Started | 2 | 1 | 0 | 1
Completed | 2 | 1 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 0 | 1 | 4
Age, Customized [Count of Participants; unit: Participants]
  8-20 years | 2 | 1 | 0 | 1 | 4
Gender [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 0 | 2
  Male | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 |  | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity
Description: A total of 7 patients enrolled on the trial. However, 2 participants withdrew from the trial before they were randomized and 1 participant withdrew from the trial before being treated. Hence, the total number of patients for assessment is 4.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Placebo
Number analyzed (Participants) | 2 | 1 | 0 | 1
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketamine 0.25 mg/kg/Dose | Ketamine 0.5 mg/kg/Dose | Ketamine 1 mg/kg/Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No